CLINICAL TRIAL: NCT00643643
Title: A Randomised, Double Blind, Placebo-Controlled, Multicentre Study Of UK-427,857 25mg O.D. , 50mg B.I.D., 100mg B.I.D And 300mg B.I.D. In Asymptomatic HIV Infected Patients To Investigate Pharmacodynamics, Pharmacokinetics, Safety And Toleration.
Brief Title: Pharmacokinetics, Pharmacodynamics, And Safety Of Maraviroc (UK-427,857) In Patients With Human Immunodeficiency Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A4001007
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Naïve
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857)
- B (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857)
- C (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857)
- D (Experimental)
  Interventions: Drug: Maraviroc (UK-427,857)
- E (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Maraviroc (UK-427,857) — 25 mg oral tablet once daily for 10 days
  Other Names: Celsentri, Selzentry
  Arms: A
Drug: Maraviroc (UK-427,857) — 50 mg oral tablet twice daily for 10 days
  Other Names: Celsentri, Selzentry
  Arms: B
Drug: Maraviroc (UK-427,857) — 100 mg oral tablet twice daily for 10 days
  Other Names: Celsentri, Selzentry
  Arms: C
Drug: Maraviroc (UK-427,857) — 300 mg oral tablet twice daily for 10 days
  Other Names: Celsentri, Selzentry
  Arms: D
Other: Placebo — Matching placebo oral tablet twice daily for 10 days
  Other Names: Celsentri, Selzentry
  Arms: E

SUMMARY:
To investigate the relationship between the pharmacokinetics and pharmacodynamics of UK-427,857 and its antiviral effects in patients with human immunodeficiency virus (HIV).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Male with HIV or surgically sterilized female with HIV showing no symptoms of HIV
* Weight between 50 and 90kg and within the permitted range for their height

Exclusion Criteria:

Exclusion criteria:

* Subjects with a CD4 count less than 250cells/mm3 or HIV viral load of less than 5000 copies/mL
* Subjects with acquired immune deficiency syndrome (AIDS) or a previous AIDS diagnosis
* Subjects whose HIV infection has been diagnosed less than 3 months prior to screening, or for who there is evidence of recent seroconversion
* Subjects who have taken anti-retroviral drugs in the eight weeks prior to the study screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2002-10; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in viral load | Day 11
Pharmacokinetic profile of UK-427,857 | Days 1 and 10
Receptor saturation | Days 1, 5, 10, 11, 13, 15, 19, 40

SECONDARY OUTCOMES:
12-lead electrocardiography | Days 1-11 and Day 40
Time course of viral load from baseline to follow-up | Days 1-15 and Days 19, 22, 25, 40
Time to rebound of viral load | Days 1-15 and Days 19, 22, 25, 40
The relationship of change in viral load (from baseline to day 11) versus average (Days 1-11) and trough (Day 10) plasma concentrations | Days 1-11
The relationship of change in viral load (from baseline to day 11) versus mean receptor saturation (Day 10) | Days 1-11
The relationship of change from baseline in viral load versus baseline virus susceptibility (IC 50 and IC 90) | Days 1-11
Adverse events | Days 1-40
Laboratory safety testing | Days 1, 3, 7, 11, 15, 40
Physical examination | Days 1, 11, 40
Supine and standing blood pressure and pulse rate | Days 1-11 and Day 40

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Germany (3):
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, München
- Pfizer Investigational Site, Utrecht, Netherlands
- Pfizer Investigational Site, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001007&StudyName=Pharmacokinetics%2C%20Pharmacodynamics%2C%20And%20Safety%20Of%20Maraviroc%20%28UK-427%2C857%29%20In%20Patients%20With%20Human%20Immunodeficiency%20Virus